CLINICAL TRIAL: NCT00812071
Title: Phase 1 Study of the Safety and Immunogenicity of RiVax With Alum in Healthy Adults
Brief Title: Phase 1B Study of RiVax, a Vaccine to Prevent the Toxic Effects of Ricin
Acronym: FDA-OPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ellen Vitetta, Director, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3369-01; 1R01FD003369-01A1 (FDA)
Record Dates: First submitted 2008-12-15; First posted 2008-12-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — RiVax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: RiVax — vaccine

SUMMARY:
Dose escalation study: 3 dose groups. 5 patients in each dose group, then 15 more patients in "best" group. 3 vaccinations in volunteers, at 0 6 and 16 weeks.

DETAILED DESCRIPTION:
Final report was submitted to Dr. Karen Russell at FDA, Rockville on September 26, 2012.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged 18-31, m or f

Exclusion Criteria:

* immunodeficiency
* pregnant
* chronic disease
* parental IgG
* abnormal labs
* drug use
* hiv
* hep c
* hep b

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
assess the safety of 3 dose levels | one year

SECONDARY OUTCOMES:
determine the immunogenicity of the 3 dose levels | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lubin, Dr., Principal Investigator — Lubin Clinic
Locations (1):
- Hampton Roads Center For Clinical Research, Chesapeake, Virginia, United States